CLINICAL TRIAL: NCT06810531
Title: Comparison Between Intravenous Ondanosteron and Metclopromide Versus Ondanesteron and Dexamethasone Effects on the Prevention of Postoperative Nausea and Vomiting in Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aiman Al-Touny (Other)
Responsible Party: Sponsor-Investigator, Aiman Al-Touny, Lecturer of Anesthesia and Intensive Care, Suez Canal University
Organization: Suez Canal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4959#
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV; IONV; cesarean section; dexamethasone; metoclopramide; Ondanesterone
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group D (Ondanesterone plus dexamethasone) (Active Comparator): patients allocated in this group will receive 4mg Ondanesterone plus 8 mg dexamethasone slowly intravenous 15 minutes before spinal anesthesia.
  Interventions: Drug: Ondanesterone plus dexamethasone combination
- Group M (ondanesterone plus metoclopramide) (Active Comparator): patients allocated in this group will receive 4mg Ondanesterone plus 10 mg metoclopramide slowly intravenous 15 minutes before spinal anesthesia.
  Interventions: Drug: ondanesterone plus metoclopramide combination

INTERVENTIONS:
Drug: Ondanesterone plus dexamethasone combination — Group D: Ondanesterone 4mg plus dexamethasone 8mg All the drugs will be prepared and diluted by normal saline in 10 ml syringe by an anesthesiologist who is not included in the study.
  The drugs will be slowly injected intravenous 15 minute from spinal anesthesia.
  Arms: Group D (Ondanesterone plus dexamethasone)
Drug: ondanesterone plus metoclopramide combination — Group M: ondanesterone 4mg plus metoclopramide 10 mg All the drugs will be prepared and diluted by normal saline in 10 ml syringe by an anesthesiologist who is not included in the study.
  The drugs will be slowly injected intravenous 15 minute from spinal anesthesia.
  Arms: Group M (ondanesterone plus metoclopramide)

SUMMARY:
The goal of this clinical trial is to prevent intraoperative nausea and vomiting (IONV) and postoperative nausea and vomiting (PONV) through comparing the efficacy of combination ondanosteron plus metclopromide versus ondanesteron plus dexamethasonein in cesarean section . The main objective is to compare the incidence of PONV between the two groups in the first 24 hours.

Patients will be randamized allocated into two groups: Group D (Ondanesterone plus dexamethasone) or Group M (ondanesterone plus metoclopramide) .

DETAILED DESCRIPTION:
Introduction Cesarean section considered one of the most surgical interventions worldwide about 7%. About 80% of pregnant women suffer from Intra and postoperative nausea and vomiting (IONV and PONV) during cesarean delivery under spinal anesthesia.

IONV and PONV decrease patients' satisfaction, increase hospital stay and can lead to wound dehiscence, bleeding, water and electrolyte abnormalities, and rehospitalization. Majority of patients prefer to experience postoperative pain rather than nausea and vomiting.

Many causes may trigger IONV and PONV and most of them are preventable. Causes of IONV may be classified into anesthetic and surgical factors. Anesthetic factors such as hypotension due to spinal anesthesia and use of some drugs like utertonics, antibiotics and opioids. Surgical factors as visceral stimulation and uterine exteriorization. PONV is mainly triggered by the emetogenic effects of opioids and severe pain.

The National Institute for Health and Care Excellence (NICE) guidelines and Enhanced Recovery after Cesarean delivery (ERAC) protocols recommend prophylactic antiemetic therapy.

Ondanesteron (5HT3 receptor antagonists) alone or with combination considered the gold standard for prophylaxis of intra and post operative nausea and vomiting.

Metoclopramide (Dopaminergic antagonists) is effective in preventing IONV more than PONV in women undergoing cesarean delivery while Dexamethasone is more appropriate for PONV due to its delayed onset.

Obstetric patients are considered high-risk group for IONV and PONV for whom combination antiemetic therapy are recommended. Till now there is no definite recommendation for best effective combination for prevention of IONV and PONV.

We aim to compare Ondanesteron plus Metchlopromide versus ondanesterone plus dexamethasone for prevention of both IONV and PONV in cesearean delivery.

Aim of Work To improve the patients' recovery and satisfaction after cesarean section, by preventing IONV and PONV through comparing the efficacy of combination ondanosteron plus metclopromide versus ondanesteron plus dexamethasone.

Sample size justification

N = (Zα/2+Zβ)2 * (p1(1-p1)+p2(1-p2)) / (p1-p2)2

Where Zα/2 = 1.96 for a confidence level of 95% Zβ = 1.64 for a power of 95% P1 = 65.6 the expected proportions of the PONV in the first 24 hours among group with metoclopramide.

P2 = 31.3 the expected proportions of the PONV in the first 24 hours among group with dexamesthsone.

Sample size by the equation will be 49 patients. And after adding 10% for drop out the sample size will be 54 patients per group.

Study population

Randomization:

Patients will be allocated into two groups: Group D (Ondanesterone plus dexamethasone) (n=54), Group M (ondanesterone plus metoclopramide) (n=54). Randomization will be carried out by a computer-generated list of random numbers, which will be sealed in an opaque envelope.

Before anesthesia, an anesthesiologist who is not included in the study will open the sealed envelope and prepare the study drugs in two 10ml syringes to be given slowly intravenous 15 minutes before the spinal anesthesia.

Patients will be recruited according to the following inclusion and exclusion criteria.

Methods:

After standard ASA monitoring, 18 G intravenous cannula will be inserted and coload with 10 ml/Kg ringer solution will be started. After that the coded study medications will be given 15 minutes before spinal anesthesia.

Spinal anesthesia will be done using 25 G quincke spinal needle. 12.5 mg heavy bupivacaine plus 100 mcg morphine will be injected intrathecal in L3-4 / L4-5 intervertebral space. All patients lying in 15 degree left lateral position and the sensory block level will be kept at T4 dermatome to decrease the risk of intra operative hypotension and provide adequate anesthestic level. Ephedrine 6 mg will be given I.V immediately after S.A to avoid intraoperative hypotension. Intraoperative hypotension (>20% from baseline) will be managed by incremental doses of 10 mg Ephedrine. After fetus delivery oxytocin 5 IU will be given slowly.

Outcome Measures Hemodynamic parameters such as heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP) and mean blood pressure (MBP) will be recorded at the following time points: baseline, every 5 minutes after spinal anesthesia administration in the first 20 minutes, then every 10 minutes till the end of the operation, in post anesthesia care unit (PACU) and every 6 hours in the ward for 24 hours postoperative.

Nausea is defined as a subjectively unpleasant sensation associated with the urge to vomit. Incidences of vomiting include retching (defined as the labored, spastic, rhythmic contraction of the respiratory muscles without expulsion of the gastric contents) and actual vomiting (defined as the forceful expulsion of gastric contents from the mouth).

Nausea and vomiting will be evaluated by means of Bellville scoring score (0: no symptoms, 1: nausea 2: retching 3: vomiting). In presence of nausea; its severity will be assessed by numeric rating scale (NRS); circling a number between "0" (labeled "no nausea") and "10" (labeled "unbearable nausea"), with unit change to left or right recorded as negative or positive, respectively.

Patients will be treated with 1 mg of Granisetron I.V in case of nausea NRS >7 and/or one emesis episode. If the emesis occurred again after 30 minutes from giving Granisetron, another 1 mg will be used till a maximum dose of 3 mg/ day The incidence of nausea and vomiting will be recorded intraoperative and postoperative during the assessment periods at 6, 12, 18, and 24 h after surgery.

Secondary Outcomes

The secondary outcomes include the following:

1. Other adverse reactions induced by the drugs, which include the following: (a) flush, (b) diarrhea, (c) headache, (d) elevated blood pressure, (e) chest congestion (f) tremors stiff muscles (g) involuntary facial movement.
2. The patient satisfaction: the patients will complete a simple questionnaire (0, very satisfied; 1, satisfied; 2, not satisfied) while they leave the PACU.
3. Post operatively pain severity will be assessed by using visual analogue scale (VAS) during follow-up visits in the PACU & ward. The VAS is a unidirectional measure of the intensity of pain. It is composed of a horizontal scale, 10 cm in length. It is anchored by two verbal pain extremes. An extreme was represented by "no pain" (scored as 0) and the other extreme was represented by "the worst pain ever" (scored as 10). The patients were told to place a mark on the scale that represents the extent of pain they suffer. The score was determined by measuring the distance between the "no pain" extreme and the mark determined by the patient. This gave a range of scores from 0- 100. A higher score indicated a severe pain. If VAS score pain is above 3 points 4 mg/kg nalbuphin will be given.
4. Time to first antiemetic need will be recorded.
5. total dose of antiemetic given in the first 24 hours after delivery will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. ASA II and III pregnant patients scheduled for elective C.S under spinal anesthesia
2. Age 18-45 years
3. Fasting before the procedure for 8 hours from solid food intake and 2 hours from water intake

Exclusion Criteria:

1. Patients with ASA physical status > III.
2. BMI >40.
3. History of motion sickness and extrapyramidal disease.
4. Smokers.
5. History of allergy to any of involved drugs in the study.
6. Patients developed nausea and vomiting and/or received antiemetic drugs within 24 hours prior to surgery.
7. History of hyperemesis gravidarum.
8. History of peptic ulcer disease.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant females scheduled for cesarean section
Enrollment: 108 (Actual)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
incidence of PONV | The first 24 hours postoperative
  Comparing the incidence of PONV between the two groups in the first 24 hours between the two groups

SECONDARY OUTCOMES:
Incidence of IONV | During the surgery
  Comparing the incidence of IONV between the two groups during the surgery.
Intraoperative non invasive blood pressure | every 5 minutes for the first 20 minutes then every 10 minutes (with a maximum of 60 minutes)during the surgery
  Intraoperative non invasive blood pressure (mmHg) changes between the two groups
Rescue antiemetic | Intraoperaotive till 24 hours postoperative
  Compare the duration needed for the first request of rescue antiemetic in minutes.
Total antiemetic dose | The first 24 hours postoperative
  Total antiemetic dose will be used in the first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Aiman Al-Touny, MD, Principal Investigator — Suez Canal University; Abdelrahman Mahmoud, MD, Principal Investigator — Suez Canal University
Locations (1):
- Suez Canal University Hospitals, Ismailia, Ismailia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 18 months following article publication.
Access Criteria: by email